CLINICAL TRIAL: NCT07140094
Title: Long-Covid-19 Alleviation Through Learning Mindfulness Study (LONG-CALM)
Brief Title: Long-Covid-19 Alleviation Through Learning Mindfulness Study
Acronym: LONG-CALM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Deborah A. Theodore, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAT0564
Record Dates: First submitted 2025-08-21; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Long COVID; Long Covid19; Post-Acute COVID-19; Post-Acute COVID-19 Syndrome; Post-Acute COVID-19 Infection; COVID Long-Haul
Keywords: Covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Receives Mindfulness Based Intervention (MBI) Immediately (Other): Group 1 participants will receive the study mindfulness intervention at the beginning of the study, along with their regular treatment as usual (through their medical providers)
  Interventions: Behavioral: Structured mindfulness intervention
- Group 2 - Receives Intervention with 8-week Delay (Other): Group 2 will begin the study with treatment as usual; they will receive the study mindfulness intervention two months after study enrollment.
  Interventions: Behavioral: Structured mindfulness intervention

INTERVENTIONS:
Behavioral: Structured mindfulness intervention — The mindfulness intervention is a series of recorded mindfulness sessions, which were created by the study team. The mindfulness recordings are between two and twenty minutes long and are accessed online.

SUMMARY:
This research is being done to study a mindfulness intervention among people who have symptoms of Post-Acute Sequelae of SARS-CoV-2 infection (PASC), also known as Long COVID. Mindfulness is defined as paying attention to the present moment with non-judgment and acceptance. Here the investigators are studying whether a mindfulness intervention can help reduce stress, reduce Long COVID symptoms, and improve quality of life among people living with Long COVID. The mindfulness intervention is a series of recorded mindfulness sessions, which were created by the study team. People who decide to take part will be randomly assigned to receive the study mindfulness intervention immediately after joining the study or to receive the study mindfulness intervention 8 weeks after joining the study. All participants will continue their usual medical care. Participants will complete online surveys to measure symptoms over time. The study will last 6 months.

DETAILED DESCRIPTION:
Patients with COVID-19 disease who go on to develop Post-Acute Sequelae of SARS-CoV-2 infection (PASC) are under significant physical and psychosocial stress. Mindfulness, operationally defined as paying attention to the present moment with non-judgment and acceptance, is a candidate treatment to reduce stress in patients with PASC. Reducing stress is critical, as stress may trigger flares in PASC symptoms. Mindfulness-Based Interventions (MBIs), including Mindfulness-Based Stress Reduction, have been shown in clinical trials, and confirmed in meta-analytic studies, to improve physical and psychological indices of stress in a wide variety of clinical and non-clinical populations. Such studies suggest an MBI might be feasible and acceptable for patients with PASC and may improve PASC symptoms and quality of life. The investigator proposes to test whether an MBI among patients with PASC alleviates symptoms.

The MBI is an 8-week online intervention that consists of a series of recorded mindfulness sessions that were developed specifically for people with PASC. The goal of the MBI is to reduce stress, reduce symptoms of PASC, and improve quality of life. Symptoms are assessed through the completion of online surveys (four surveys over 6 months). All participation is remote (no in-person study visits).

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18
* Willing and able to provide informed consent
* Access to the internet
* Self-reported history of SARS-CoV-2 infection
* Current symptoms attributed to PASC by participant or by participant's medical provider; ongoing symptoms that persisted >= 12 weeks after Covid-19 illness

Exclusion Criteria:

* Participating in another clinical trial of an intervention for PASC symptoms
* Engaged in a structured MBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-05-21 (Estimated); Study Completion 2027-11-21 (Estimated)

PRIMARY OUTCOMES:
Mean Score of Patient-Reported Outcomes Measurement Information System (PROMIS) Global 10 Score | Month 2
  This is to compare the difference between both groups at Month 2. The PROMIS Global 10 is a health-related quality of life measure. Raw scores range from 4 to 20. A higher score indicates better health.

SECONDARY OUTCOMES:
Change in PROMIS Global 10 Score | Months 1, 2, 6
  The PROMIS Global 10 is a health-related quality of life measure. Raw scores range from 4 to 20. A higher score indicates better health.
Post-Acute Sequelae of SARS-CoV-2 (PASC) Score | Months 1, 2, 6
  This study uses the PASC score defined by Thaweethai et al., JAMA, 2023. The PASC score is measured as the sum of the scores for each PASC symptom reported by a participant at the specified timepoint. See: doi:10.1001/jama.2023.8823.
Patient Health Questionnaire 9 (PHQ9) Score | Months 1, 2, 6
  The PHQ9 is a 9-item questionnaire measuring depression symptoms. The scores range from 0 to 27, with higher scores indicating greater severity.
Generalized Anxiety Disorder 7 (GAD7) Score | Months 1, 2, 6
  The GAD7 is a 7-item scale that measures anxiety symptoms. The scores range from 0 to 21, with higher scores indicating greater severity.
Impact of Event 6 (IES-6) Scores | Months 1, 2, 6
  IES-6 is a 6-item scale that measures post traumatic stress disorder (PTSD) symptoms. The scores range from 0 to 18, with higher scores indicating greater severity.
State Mindfulness Scale for Physical Activity Score | Months 1, 2, 6
  The State Mindfulness Scale for Physical Activity Score measures mindfulness after physical activity. There are twelve questions, each scored between 0-4. The scores for each question are summed and then divided by 12. A higher score indicates a greater degree of mindfulness.
Difference in Patient-Reported Outcomes Measurement Information System (PROMIS) Global 10 Score | Months 1 and 6
  Mean score difference in health-related quality of life, as measured by PROMIS Global 10 criteria. The PROMIS Global 10 is a health-related quality of life measure. Raw scores range from 4 to 20. A higher score indicates better health.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Theodore, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thaweethai T, Jolley SE, Karlson EW, Levitan EB, Levy B, McComsey GA, McCorkell L, Nadkarni GN, Parthasarathy S, Singh U, Walker TA, Selvaggi CA, Shinnick DJ, Schulte CCM, Atchley-Challenner R, Alba GA, Alicic R, Altman N, Anglin K, Argueta U, Ashktorab H, Baslet G, Bassett IV, Bateman L, Bedi B, Bhattacharyya S, Bind MA, Blomkalns AL, Bonilla H, Brim H, Bush PA, Castro M, Chan J, Charney AW, Chen P, Chibnik LB, Chu HY, Clifton RG, Costantine MM, Cribbs SK, Davila Nieves SI, Deeks SG, Duven A, Emery IF, Erdmann N, Erlandson KM, Ernst KC, Farah-Abraham R, Farner CE, Feuerriegel EM, Fleurimont J, Fonseca V, Franko N, Gainer V, Gander JC, Gardner EM, Geng LN, Gibson KS, Go M, Goldman JD, Grebe H, Greenway FL, Habli M, Hafner J, Han JE, Hanson KA, Heath J, Hernandez C, Hess R, Hodder SL, Hoffman MK, Hoover SE, Huang B, Hughes BL, Jagannathan P, John J, Jordan MR, Katz SD, Kaufman ES, Kelly JD, Kelly SW, Kemp MM, Kirwan JP, Klein JD, Knox KS, Krishnan JA, Kumar A, Laiyemo AO, Lambert AA, Lanca M, Lee-Iannotti JK, Logarbo BP, Longo MT, Luciano CA, Lutrick K, Maley JH, Mallett G, Marathe JG, Marconi V, Marshall GD, Martin CF, Matusov Y, Mehari A, Mendez-Figueroa H, Mermelstein R, Metz TD, Morse R, Mosier J, Mouchati C, Mullington J, Murphy SN, Neuman RB, Nikolich JZ, Ofotokun I, Ojemakinde E, Palatnik A, Palomares K, Parimon T, Parry S, Patterson JE, Patterson TF, Patzer RE, Peluso MJ, Pemu P, Pettker CM, Plunkett BA, Pogreba-Brown K, Poppas A, Quigley JG, Reddy U, Reece R, Reeder H, Reeves WB, Reiman EM, Rischard F, Rosand J, Rouse DJ, Ruff A, Saade G, Sandoval GJ, Santana JL, Schlater SM, Sciurba FC, Shepherd F, Sherif ZA, Simhan H, Singer NG, Skupski DW, Sowles A, Sparks JA, Sukhera FI, Taylor BS, Teunis L, Thomas RJ, Thorp JM, Thuluvath P, Ticotsky A, Tita AT, Tuttle KR, Urdaneta AE, Valdivieso D, VanWagoner TM, Vasey A, Verduzco-Gutierrez M, Wallace ZS, Ward HD, Warren DE, Weiner SJ, Welch S, Whiteheart SW, Wiley Z, Wisnivesky JP, Yee LM, Zisis S, Horwitz LI, Foulkes AS; RECOVER Consortium. Development of a Definition of Postacute Sequelae of SARS-CoV-2 Infection. JAMA. 2023 Jun 13;329(22):1934-1946. doi: 10.1001/jama.2023.8823. PMID 37278994